CLINICAL TRIAL: NCT01753869
Title: Timing of Hypertonic Saline Inhalation Relative to Airways Clearance in Cystic Fibrosis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Challenges with recruitment
Sponsor: Belfast Health and Social Care Trust (Other)
Collaborators: Queen's University, Belfast (Other); University of Ulster (Other)
Responsible Party: Principal Investigator, Katherine O'Neill, PhD researcher on behalf of PI: Prof Judy Bradley, Queen's University, Belfast
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 12025JB-AS
Record Dates: First submitted 2012-12-13; First posted 2012-12-20 (Estimated); Last update posted 2016-07-19 (Estimated); Status verified 2016-07

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ACTs after HTS inhalation: (Active Comparator): ACTs after HTS inhalation: Patients will take a bronchodilator (Salbutamol, 2 puffs) wait 15 minutes, and then take a single inhalation (4 mls) of 7% HTS (Nebusal™) via updraft nebulizer (Portex) (approximately 20 minutes) immediately followed by an airways clearance session of 10 supervised cycles of Active Cycle of Breathing Technique (ACBT) using the acapella® (approximately 20 minutes).
  Interventions: Procedure: Airways clearance and Hypertonic saline inhalation
- ACTs during HTS inhalation (Active Comparator): ACTs during HTS inhalation: Patients take a bronchodilator (Salbutamol, 2 puffs), wait 15 minutes, and then take a single inhalation (4mls) of 7% HTS (Nebusal™) through the acapella® duet (with portex updraft nebulizer attached) device. During inhalation, an airways clearance session of 10 supervised cycles of ACBT using the acapella® will be carried out (approximately 20 minutes).
  Interventions: Procedure: Airways clearance and Hypertonic saline inhalation

INTERVENTIONS:
Procedure: Airways clearance and Hypertonic saline inhalation

SUMMARY:
Lung disease is the predominant cause of morbidity and mortality in Cystic Fibrosis (CF) with 80% of deaths resulting directly or indirectly from pulmonary disease. Abnormal airway clearance causes retention of mucus resulting in frequent chest infections. Physiotherapists use different techniques to help clear mucus from the lungs of patients with CF. Inhaled medications and airways clearance techniques (ACTs) are central to a CF patient's daily treatment and are often coordinated.

Burden of treatment is a common reason for non-adherence in this patient group, and streamlining of treatment timings is sought to optimize adherence whilst ensuring efficacy to an often complex daily regimen of inhaled bronchodilators, nebulizers and ACTs. A gap in the research exists as to the optimal timing of Hypertonic Saline (HTS) and ACT within the daily regimen. A study to show whether the timing of HTS around ACT is significant, can better inform patients and potentially allow more flexibility around their treatment regimen.

Lung Clearance Index (LCI) has shown good sensitivity to abnormalities in lung function compared with spirometry and has demonstrated a treatment effect in other trials. LCI may be a suitable tool therefore, to assess intervention strategies aimed at airways clearance in CF. This study aims to compare the effects ACTs after HTS inhalation versus ACTs during HTS inhalation as measured by LCI.

It is a randomized, crossover trial of ACTs after HTS inhalation compared with ACTs during HTS inhalation in adult CF patients during day 10-14 of a hospital admission for treatment of a pulmonary exacerbation. Patients will be randomized to receive 1 of the treatment session options on the first day and the reverse on the second day.

The primary objective of this study is to compare the change in LCI (a measure of lung function) at 90 minutes post treatment with ACTs after HTS inhalation compared with ACTs during HTS inhalation in adult CF patients.

LCI (lung clearance index) ACT (airway clearance technique) HTS (hypertonic saline)

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients with a documented diagnosis of CF aged ≥18 years.
2. Written informed consent.
3. At least day 10 - 14 of IV antibiotic therapy during a hospital admission for a pulmonary exacerbation.
4. Patients must be able to perform acceptable spirometric manoeuvres, according to the American Thoracic Society/ERS (ATS/ERS) standards (Miller, Hankinson et. al. 2005).
5. Patient with an FEV1% predicted of ≥ 40%predicted (Stanojevic, Wade et al. 2008).
6. Patients who are productive of sputum from screening visit to study visit 1 (≥10g over 24 hours).
7. Patients who have been prescribed HTS (Nebusal 7%) and have successfully completed a challenge test.
8. Any other chronic medication must have commenced therapy 4 weeks prior to screening and be willing to continue this therapy for the entire duration of the study.

Exclusion Criteria:

1. Day 1-9 of IV antibiotic therapy during a hospital admission.
2. Patients who are colonized with Burkholderia cepacia complex.
3. Patient who are HTS naive.
4. Patients who have an intolerance to HTS.
5. Patients who are currently participating in another study or have participated in another study with an investigational drug within one month of screening.
6. Clinically significant disease or medical condition other than CF or CF-related conditions that, in the opinion of the Investigator, would compromise the safety of the patient or the quality of the data.

   -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2012-12; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Lung Clearance Index | 90 minutes post treatment

SECONDARY OUTCOMES:
24 hour sputum volume | 24 hours post treatment

OTHER OUTCOMES:
spirometry (FEV1% predicted; FEF25-75% [Forced expiratory flow 25-75] predicted) | 90 minutes post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Judy M Bradley, PhD, Principal Investigator — University of Ulster
Locations (1):
- Belfast Health and Social Care Trust, Belfast City Hospital, Belfast, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Morrison L, Milroy S. Oscillating devices for airway clearance in people with cystic fibrosis. Cochrane Database Syst Rev. 2020 Apr 30;4(4):CD006842. doi: 10.1002/14651858.CD006842.pub5. PMID 32352564
- [Derived] O'Neill K, Moran F, Tunney MM, Elborn JS, Bradbury I, Downey DG, Rendall J, Bradley JM. Timing of hypertonic saline and airway clearance techniques in adults with cystic fibrosis during pulmonary exacerbation: pilot data from a randomised crossover study. BMJ Open Respir Res. 2017 Jan 12;4(1):e000168. doi: 10.1136/bmjresp-2016-000168. eCollection 2017. PMID 28123751